CLINICAL TRIAL: NCT00146341
Title: An Eight Week Randomized, Double-Blind, Double-Dummy Study Comparing a Fixed Dose Combination of Telmisartan 80mg Plus Hydrochlorothiazide 12.5mg to Telmisartan 80mg in Patients Who Fail to Respond Adequately to Treatment With Telmisartan 80mg.
Brief Title: Combination of Telmisartan 80 mg Plus Hydrochlorothiazide 12.5 mg to Telmisartan 80 mg in Patients Failed in Telmisartan 80 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.472
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

INTERVENTIONS:
Drug: Telmisartan/HCTZ
Drug: Telmisartan

SUMMARY:
To demonstrate that a fixed dose combination of telmisartan 80 mg plus HCTZ 12.5 mg is superior to telmisartan 80 mg alone in patients, who fail to respond adequately to telmisartan 80 mg monotherapy, in lowering seated trough diastolic blood pressure after eight weeks of treatment.

DETAILED DESCRIPTION:
This is a multi-centre, prospective, randomized, double-blind, parallel-group study in approximately 244 patients with a history of mild-to-moderate hypertensive who have been shown not to respond to telmisartan monotherapy.

All patients will enter a one-week screening phase prior to starting the eight-week open-label T80 mg period. At the end of four weeks, only patients who fail to respond to T80 mg (DBP >= 90 mm Hg) will continue the treatment with T80 mg for another four weeks. At the end of eight weeks, only patients who fail to respond to T80 mg (DBP >= 90 mm Hg) will be randomized, double-blind, to receive either T80 mg alone or the fixed dose combination of T80 mg plus HCTZ 12.5 mg for eight weeks. Seated BP will be taken 24 hours post-dose at each visit. Labs, ECG, and physical examination will be done at screening, at baseline and at the final visit.

Study Hypothesis:

The primary objective of the study, showing that fixed dose combination is superior to telmisartan 80 mg alone will be tested using the hypotheses given below.

H0: u T80/H12.5 - uT80 = 0 mm Hg versus H1: uT80/H12.5 - uT80 not equal 0 mm Hg, where uT80/H12.5 anduT80 represent the average reduction from baseline (Visit 4) in trough seated DBP for the fixed dose combination and telmisartan 80 mg, respectively.

Testing of the null hypothesis will be performed using a two-sided test of significance at an a-level (type-I error rate) of 0.05.

Comparison(s):

The primary efficacy endpoint will be the change from baseline in seated DBP 24 hours post-dose at the last visit during the double-blind treatment phase. The pre-dose measurement on visit 4 will be viewed as the baseline measurement.

ELIGIBILITY:
Inclusion Criteria:

1. History of mild-to-moderate hypertension defined by a mean seated DBP >=95 and <= 109 mmHg before inclusion in the open-label phase
2. Patients who fail to respond adequately to telmisartan monotherapy (mean seated DBP >= 90 mmHg)
3. Participants between 18 and 80 years of age
4. Ability to provide written informed consent

Exclusion Criteria:

1. Patients taking more than three anti-hypertensive medications at the screening visit.
2. Pre-menopausal women (last menstruation 1 year prior to start of screening):

   * Who are not surgically sterile (hysterectomy, tubal ligation)
   * Who are NOT practicing acceptable means of birth control or who do NOT plan to continue using an acceptable method throughout the study (acceptable methods of birth control include IUD, oral, implantable or injectable contraceptives)
3. Any woman:

   * Who has a positive urine pregnancy test at screening (Visit 1)
   * Who is nursing
4. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   * SGPT(ALT) or SGOT(AST) greater than two times the upper limit of normal
   * Serum creatinine > 3.0 mg/dL (or 265 mol/L) or creatinine clearance < 0.6 ml/sec
5. Clinically relevant hypokalaemia or hyperkalaemia
6. Uncorrected volume depletion
7. Uncorrected sodium depletion
8. Primary aldosteronism
9. Hereditary fructose intolerance
10. Biliary obstructive disorders, cholestasis or moderate to severe hepatic insufficiency
11. Known or suspected secondary hypertension
12. Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney
13. Congestive heart failure (NYHA functional class CHF III-IV)
14. Unstable angina within the past three months
15. Stroke within the past six months
16. Myocardial infarction or cardiac surgery within the past three months
17. PTCA within the past three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2005-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09

PRIMARY OUTCOMES:
The primary efficacy variable is change from baseline in seated DBP at trough (24 hours post-dosing) after eight weeks of randomized treatment or at last trough observation during the double-blind phase (i.e. last trough observation carried forward).

SECONDARY OUTCOMES:
Change from baseline in seated SBP, standing DBP and SBP at trough after eight weeks of randomized treatment or at last trough observation during the double-blind phase. The percentage of patients responding to the treatment. Safety.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (9):
- China (9):
  - China-Japan Friendship Hospital, Beijing
  - Beijing Tiantan Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - No. 1 Hospital Affiliated Nanjing, Nanjing
  - Ruijin Hospital, School of Medicine, Shanghai
  - Shanghai Changhai Hospital, Shanghai
  - 254 PLA Hospital, Tianjin
  - Second Hospital Affiliated to Tianjin Med University, Tianjin
  - No. 1 Hosp Affiliated to Med College, Zhejiang Province

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24493330